CLINICAL TRIAL: NCT00000406
Title: Effects of Strength Training on Knee Osteoarthritis (OA)
Brief Title: Effects of Strength Training on Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: P60 AR20582 Substudy EEHSR3; P60AR020582 (NIH); NIAMS-022
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis (OA); Knee; Radiographic OA; Strength training; Physical therapy; Exercise; Body composition; Striated muscle; Depression; Radiographic OA with knee pain; Radiographic OA without knee pain; Knee pain without radiographic OA; Normal elderly (no radiographic OA, no knee pain)
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity; Depression

INTERVENTIONS:
Procedure: Progressive resistance exercise

SUMMARY:
To understand the effects of leg strengthening exercise, we will study the effects of strength training of the legs in four groups of people: (1) osteoarthritis (OA) with knee pain; (2) OA without knee pain; (3) no OA but elderly with knee pain; and (4) normal elderly with no OA or knee pain. In each of the first three groups, we will look at whether people who do strength training have less pain and/or slower progression of x-ray signs of OA over 30 months than people who perform nonstrengthening, range-of-motion exercises. We are including the fourth group to find out whether people with OA (groups 1 & 2) have the same response to strength training as healthy elderly people, and whether those with knee pain (groups 1 & 3) have the same response to training as those without joint pain.

DETAILED DESCRIPTION:
Several studies have confirmed that weak leg muscles are associated with osteoarthritis (OA) of the knee. Studies of body composition in these people have also shown that, despite being weaker, people with OA have significantly greater muscle mass than those without OA, suggesting that those with OA may have the potential to greatly increase their strength. However, research has not clearly shown whether exercises designed to improve leg strength will decrease the severity of pain or slow the progression of OA based on radiographic (x-ray) analysis. To understand the effects of leg strengthening exercise, we will perform a randomized clinical trial of lower extremity strength training using four subgroups of people: (1) OA with knee pain; (2) OA without knee pain; (3) no OA with knee pain; and (4) normal elderly with no OA or knee pain.

In each of the first three groups, we will determine whether people assigned to strength training have lower pain scores and/or slower progression of radiographic changes of OA over 30 months than controls who perform nonstrengthening exercises (i.e., range-of-motion exercises). We are including the fourth group to determine whether those with OA (groups 1 & 2) exhibit the same response to strength training as healthy elderly people, and whether those with knee pain (groups 1 & 3) have the same response to training as those without joint pain. We will also prospectively monitor changes in body composition and bone mass, quality of life, and symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 60 to 100 years of age

Exclusion Criteria:

* Knee joint replacement surgery
* Diabetes mellitus
* Uncontrollable hypertension
* Neuropathies of the lower extremity
* Poor mental cognition (i.e., inability to follow instructions)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 1977-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Mikesky, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- National Institute for Fitness and Sport, Indianapolis, Indiana, United States

REFERENCES:
- [Result] Mikesky AE, Mazzuca SA, Brandt KD, Perkins SM, Damush T, Lane KA. Effects of strength training on the incidence and progression of knee osteoarthritis. Arthritis Rheum. 2006 Oct 15;55(5):690-9. doi: 10.1002/art.22245. PMID 17013851